CLINICAL TRIAL: NCT03842930
Title: Embolization of the Lumbar Arteries Before EVAR: A Prospectively Randomized Trial Comparing Platinum-Fibered Microcoils (Control Arm) With the MVP® Microvascular Plug (Study Arm)
Brief Title: ELECT Trial - Embolization of the Lumbar Arteries Before EVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dierk Scheinert, Principal Investigator, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP_18/002
Record Dates: First submitted 2019-01-21; First posted 2019-02-15 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platinum-fibered Microcoils (FPC) (Other): Embolization using platinum fibred Coils (Cook Incorporated, Bloomington, IN, USA)
  Interventions: Procedure: Endovascular embolization
- MVP® Vascular Plug (Other): Embolization using MVP®-Plug (Medtronic Inc., Minneapolis, MI, USA).
  Interventions: Procedure: Endovascular embolization

INTERVENTIONS:
Procedure: Endovascular embolization — Endovascular embolization of the Lumbar Arteries

SUMMARY:
Prospective, Randomized, Single-center Study for the Treatment of Subjects with Abdominal Aortic Aneurysm: Embolization of the Lumbar Arteries Before EVAR: A Prospectively Randomized Trial Comparing Platinum-Fibered Microcoils (control arm) with the MVP® Microvascular Plug (study arm)"

DETAILED DESCRIPTION:
This study is a prospective, single-center, 1:1 randomized trial to investigate the difference in radiation dose and intervention time between the embolization with FCP and MVP-Plug.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18
2. Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved consent form.
3. Indication for the occlusion of lumbar arteries due to:

   1. Subject has an abdominal aortic aneurysm and
   2. At least 2 patent lumbar arteries in the diseased area
4. Subject understands the duration of the study, agrees to attend the stentgraft implantation
5. A microcatheter is successfully placed the target lumbar artery.

Exclusion Criteria:

1. Any surgical procedure or intervention performed within 30 days prior to or post index procedure
2. Aortic aneurysm requires treatment with alternative therapies such as operation
3. any other aortic pathology
4. major untreated cardio-pulmonary disease
5. life-expectancy of less than one year
6. expected lack of compliance (e.g. if the patient may not be willing to have several sessions and the following repair done)
7. pregnant or nursing women
8. impaired thyroid function, if not under stable treatment
9. women of child-bearing potential without highly effective contraceptive measures
10. Enrolled in another investigational drug, device or biologic study
11. Failure to successfully intubate an lumbar artery
12. Stroke or heart attack within 3 months prior to enrollment
13. Known allergies or sensitivity to heparin, aspirin, other anticoagulant/ antiplatelet therapies, paclitaxel or contrast media that cannot be adequately pre-treated prior to index procedure
14. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy.
15. Platelet count <100,000 mm3 or >600,000 mm3
16. Receiving dialysis or immunosuppressant therapy
17. Chronic kidney disease (serum creatinine > 2.5 mg/dL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Radiation dose for embolization of the lumbar arteries with the MVP plug or coils | through study completion, an average of 3-4 month

SECONDARY OUTCOMES:
Intervention time for embolization of the lumbar arteries with the MVP plug or coils | through study completion, an average of 3-4 month
Success in complete occlusion of the targeted lumbar artery | through study completion, an average of 3-4 month

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, Prof. Dr., Principal Investigator — University Clinic Leipzig
Locations (1):
- University Clinic Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Konert M, Schmidt A, Branzan D, Wittig T, Scheinert D, Steiner S. ELECT: prospective, randomized trial comparing microvascular plug versus platinum-fibered microcoils for embolization of aneurysm sac side branches before endovascular aortic aneurysm repair. CVIR Endovasc. 2024 May 3;7(1):42. doi: 10.1186/s42155-024-00454-6. PMID 38700601